CLINICAL TRIAL: NCT00297947
Title: A Randomized, Double-Blind, Parallel-Group, Fixed Dose, Clinical Trial of Quetiapine 600 mg/Day vs 1200 mg/Day for Patients With Treatment-Resistant Schizophrenia or Schizoaffective Disorder
Brief Title: High Dose of Quetiapine in Treating Subjects With Treatment Refractory Schizophrenia or Schizoaffective Disorder
Acronym: HDQ
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Manhattan Psychiatric Center (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Jean-Pierre Lindenmayer, Clinical Director, Manhattan Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRUSQUET0348
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; quetiapine; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 600 mg/day quetiapine (Group B) (Experimental): Patients qualifying for the Double Blind Phase will be randomly assigned to 600 mg quetiapine (Group B) daily and treated on the assigned dose in a double-blind fashion for 8 weeks
  Interventions: Drug: quetiapine
- 1200 mg/day quetiapine (Group A) (Experimental): Patients qualifying for the Double Blind Phase will be randomly assigned to high dose 1200 mg quetiapine daily (Group A) on the assigned dose in a double-blind fashion for 8 weeks
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: quetiapine — Participant will receive 1200 mg/day of quetiapine in twice daily dosing for 8 weeks.
  Other Names: Seroquel
  Arms: 1200 mg/day quetiapine (Group A)
Drug: quetiapine — Participant will receive 600 mg/day of quetiapine for 8 weeks.
  Other Names: Seroquel
  Arms: 600 mg/day quetiapine (Group B)

SUMMARY:
This study will investigate the safety and efficacy of quetiapine in sub-optimally responding patients with DSM-IV schizophrenia using a double blind, randomized 12-week trial comparing oral doses of 1200 mg/d to 600 mg/d of quetiapine.

DETAILED DESCRIPTION:
The study will be conducted at two sites: Manhattan Psychiatric Center (MPC), and the Clinical Research and Evaluation Facility at the Nathan S. Kline Institute for Psychiatric Research/Rockland Psychiatric Center (NKI). A total of 60 patients will be enrolled, 30 at each location. After a screening period of 1 week, all patients will be entering an open label, four-week quetiapine treatment period (run-in phase), during which quetiapine will be titrated to 600 mg PO daily and other adjunctive antipsychotics will be gradually tapered and discontinued. Other concomitant medications such as mood stabilizers will be maintained, if their dose has been stable for the preceding 2 months. Patients not responding to quetiapine treatment at 600 mg PO (defined as reduction of < 15% change in Positive and Negative Syndrome Scale (PANSS) total score between start of run-in to end of week 4) during the run-in phase, will be eligible to enter the double blind phase. Study baseline will be Day 7 of Week 4 of the run-in phase. Patients qualifying for the double-blind phase will be randomly assigned to either high dose 1200 mg quetiapine daily (Group A) or to 600 mg quetiapine (Group B) daily and treated on the assigned dose in a double blind fashion for 8 weeks (Week 1 through Week 8 of double blind phase). Measures of extra-pyramidal side effects, psychopathology, and safety will be conducted throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for chronic schizophrenia or schizoaffective disorder
2. Sub-optimal treatment-response
3. Total score > 60 on the Positive and Negative Syndrome Scale (PANSS) at baseline of run-in phase and again at baseline of double blind phase
4. Age 18-64 years old
5. Signed informed consent
6. Patient is in good general medical health

Exclusion criteria:

1. History of failure to respond to 400 mg/day or more of clozapine for 8 contiguous weeks
2. History of failure to respond to quetiapine treatment at dosages > 1200 mg daily for 6 contiguous weeks
3. History of quetiapine intolerance (e.g., clinically significant leukopenia or agranulocytosis, or severe dystonic reactions)
4. Significant recent history of violence or suicidal activity, which required > 4 episodes of PRN anti-agitation medication per week
5. Mental retardation
6. Depot antipsychotic within 30 days before randomization
7. Significant medical illness requiring frequent dose adjustment or medication changes

Clozapine non-responders are explicitly excluded, as they would be unlikely to show a response in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To see if mean extrapyramidal symptoms measure will change significantly from baseline to endpoint for the whole group and if the mean change in EPS measure is significantly different between quetiapine 1200mg daily group and quetiapine 600mg daily group | 8 weeks

SECONDARY OUTCOMES:
To see if treatment with quetiapine 1200 mg per day will improve total PANSS more robustly than quetiapine 600 mg per day | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Lindenmayer, MD, Principal Investigator — Manhattan Psychiatric Center; Leslie Citrome, MD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (2):
- United States (2):
  - Manhattan Psychiatric Center, New York, New York
  - Nathan Kline Institute for Psychiatric Research, Orangeburg, New York

REFERENCES:
- [Background] Citrome L, Jaffe A, Levine J, Lindenmayer JP. Dosing of quetiapine in schizophrenia: how clinical practice differs from registration studies. J Clin Psychiatry. 2005 Dec;66(12):1512-6. doi: 10.4088/jcp.v66n1203. PMID 16401150
- [Result] Lindenmayer JP, Citrome L, Khan A, Kaushik S, Kaushik S. A randomized, double-blind, parallel-group, fixed-dose, clinical trial of quetiapine at 600 versus 1200 mg/d for patients with treatment-resistant schizophrenia or schizoaffective disorder. J Clin Psychopharmacol. 2011 Apr;31(2):160-8. doi: 10.1097/JCP.0b013e31820f4fe0. PMID 21346616
- See also: Quetiapine on Wikipedia — http://en.wikipedia.org/wiki/Quetiapine
- See also: NIMH on Schizophrenia — http://www.nimh.nih.gov/health/topics/schizophrenia/index.shtml
- See also: Wikipedia on Schizophrenia — http://en.wikipedia.org/wiki/Schizophrenia